CLINICAL TRIAL: NCT05283005
Title: Alveolar Cleft Reconstruction Using Double Iliac Corticocancellous Bone Blocks Technique Versus Particulate Autogenous Spongy Bone Graft From Anterior Iliac Crest. A Randomized Clinical Trial
Brief Title: Alveolar Cleft Grafting by Double Iliac Bone Blocks Versus Iliac Spongy Bone From Anterior Iliac Crest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Louai Ahmed Rafat Mohammed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29-12-21
Record Dates: First submitted 2022-02-16; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Alveolar Cleft

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alveolar cleft patients will be treated by conventional technique (Active Comparator): Reconstruction of alveolar cleft by autogenous cancellous bone from the anterior iliac crest (gold standard technique).
  Interventions: Procedure: Grafting of the alveolar cleft
- alveolar cleft patients will be treated by double cortex technique (Experimental): Reconstruction of alveolar cleft by autogenous double iliac cortico-cancellous bone blocks from the anterior iliac crest.
  Interventions: Procedure: Grafting of the alveolar cleft

INTERVENTIONS:
Procedure: Grafting of the alveolar cleft — alveolar cleft grafting using either the conventional technique or the double cortex technique

SUMMARY:
Reconstruction of Alveolar Cleft Using Double Iliac Corticocancellous Blocks in comparison with the gold standard technique ( cancellous bone ) both from anterior iliac crest.

DETAILED DESCRIPTION:
This study will compare two techniques for the proper alveolar cleft reconstruction with adequate bone bridge formation of maximum bone quality, contour, and minimal resorption. One of them is packing autogenous particulate spongy bone from the anterior iliac crest (gold standard). While the other technique would be reconstruction of the cleft with two iliac corticocancellous bone blocks with cancellous bone in between. which benefits of the rapid revascularization and healing of cancellous bone and the strong mechanical properties of cortical bone that will aid in obtaining a proper reconstruction and form for the defect and can be applied to defects of any size.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete maxillary alveolar cleft either unilateral or bilateral at the age of mixed dentition (between 7 and 13 years old).

  * repaired cleft lip.
  * Patients with cleft lip and palate who have not undergone alveolar grafting procedure.
  * Patients with unerupted maxillary permanent canine in the cleft region.
  * Patients with medical history that did not hinder surgical intervention and have adequate proper oral hygiene.
  * Both genders males and females will be included

Exclusion Criteria:

* General contraindications to surgical intervention of the area. Patients with ill repaired cleft lip that will hinder the appropriate reconstruction of the alveolar cleft.

  * Patients with associated syndrome.
  * Patients requiring concomitant Orthognathic surgical procedure.
  * Subjected to irradiation in the head and neck area less than 1 year before surgery.
  * Untreated periodontitis.
  * Poor oral hygiene.
  * Uncontrolled diabetes.
  * Immunosuppressed or immunocompromised.
  * Treated or under treatment with intravenous amino-bisphosphonates.
  * Active infection or severe inflammation in the area intended for graft placement.
  * Patients participating in other studies, if the present protocol could not be properly followed.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-12-29 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring graft height in millimeters | 9 months
  CBCT scan analysis for measuring mean graft height in millimeters of every graft of both groups of patients immediately after surgery and compare it with CBCT scan analysis for measuring mean graft height in millimeters after 9 months of every graft for assessment of grafts height stability of both groups over 9 months.
Measuring graft width in millimeters | 9 months
  CBCT scan analysis for measuring mean graft width in millimeters of every graft of both groups of patients immediately after surgery and compare it with CBCT scan analysis for measuring mean graft width in millimeters after 9 months of every graft for assessment of grafts width stability of both groups over 9 months.

SECONDARY OUTCOMES:
Measuring graft volume in cubic millimeter | 9 months
  CBCT scan analysis for measuring graft volume in cubic millimeter of every graft of both groups of patients immediately after surgery and compare it with CBCT scan analysis for measuring graft volume in cubic millimeter after 9 months of every graft for assessment of grafts volume stability of both groups over 9 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo university, Cairo, Egypt